CLINICAL TRIAL: NCT01442870
Title: Prospective Evaluation of Clinical Safety of Combining Metformin With Anticancer Chemotherapy
Brief Title: Evaluation of Clinical Safety of Combining Metformin With Anticancer Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Metformin Anticancer + Chemo
Record Dates: First submitted 2011-09-21; First posted 2011-09-29 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin
  Interventions: Drug: Metformin
- No metformin (No Intervention): No metformin during primary endpoint assessment period (at least 3 weeks). Patients will subsequently be initiated on metformin.

INTERVENTIONS:
Drug: Metformin — Metformin
  Arms: Metformin

SUMMARY:
Metformin is a drug that is normally used to treat people with diabetes. New research has discovered that metformin may also kill cancer stem cells. These cancer stem cells make up only a small portion of a cancer, but may be responsible for resistance to chemotherapy or for causing recurrence of the cancer. Future studies are envisioned to that test the efficacy of administering metformin with chemotherapy. The purpose of this study is to assess the safety of administering metformin in combination with chemotherapy. Since chemotherapy and cancer itself both cause adverse events by themselves, this study is designed to have a run-in stage as well as a subsequent randomization to metformin or no metformin. The primary endpoint will compare the rate of dose-limiting toxicities between these two arms. After a period of 3 weeks for the primary endpoint comparison, all patients will receive metformin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented cancer; diagnosis of hepatocellular carcinoma may be made by characteristic radiographic and/or AFP findings 33;
* Intended treatment with, or currently being treated by anti-cancer chemotherapy in the adjuvant or advanced setting;
* Age 18 to 79;
* Adequate renal function (serum creatinine levels <1.5 mg/dL [males], <1.4 mg/dL [females]). If a subject does not meet these criteria, but does have an estimated creatinine clearance >= 60 ml/min using the Cockroft-Gault calculation, they will be allowed. The Cockroft-Gault formula is CrCl = (140-age) x weight(kg)÷(Cr x72), where CrCl = estimated creatinine clearance and Cr is plasma creatinine in mg/dL;
* Adequate hepatic parameters, including aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 x upper limit of normal (ULN), total bilirubin ≤ 1.5 x ULN, and alkaline phosphatase levels ≤ 2.5 x ULN;
* Must anticipate receiving at least 3 cycles (or treatment periods of at least 3-weeks) of chemotherapy;
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Current use of metformin (within 1 week of start of chemotherapy regimen to be assessed);
* Patients with type 2 diabetes are allowed, however they will be excluded if there is intent to use metformin for treatment of diabetes during the course of the study;
* Undergoing chemotherapy treatment concurrent with radiation therapy;
* Undergoing chemotherapy in a neoadjuvant setting prior to potentially curative surgery;
* Renal disease or renal dysfunction not meeting inclusion criteria;
* Significant medical conditions such as cardiovascular collapse (shock), acute myocardial infarction, septicemia, acute or chronic metabolic acidosis;
* History of, or states associated with, lactic acidosis such as shock or pulmonary insufficiency, alcoholism (acute or chronic), conditions associated with hypoxemia and pancreatitis;
* Severe dehydration;
* Clinical or laboratory evidence of hepatic disease;
* Congestive heart failure requiring pharmacologic treatment, or unstable or acute congestive heart failure;
* Known hypersensitivity to metformin hydrochloride;
* Pregnant or lactating women (serum pregnancy test will be performed for all women of child-bearing potential);
* Psychiatric illness or social situation that would limit compliance with study requirements and/or obscure results

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity when metformin is added to chemotherapy | 1 cycle (at least 3 weeks)
  The primary endpoint of the study will be to determine whether metformin can be safely added to a chemotherapy regimen that is previously well tolerated. The rate of dose limiting toxicities will be compared.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 cycle (at least 3 weeks)
  Secondary endpoints will include assessment of AEs ≥ grade 3 and Serious Adverse Events (SAEs), assessment of safety beyond the first cycle with metformin, and an exploration of metformin-chemotherapy drug interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Saif, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Saif MW, Rajagopal S, Caplain J, Grimm E, Serebrennikova O, Das M, Tsichlis PN, Martell R. A phase I delayed-start, randomized and pharmacodynamic study of metformin and chemotherapy in patients with solid tumors. Cancer Chemother Pharmacol. 2019 Dec;84(6):1323-1331. doi: 10.1007/s00280-019-03967-3. Epub 2019 Oct 3. PMID 31583436